CLINICAL TRIAL: NCT04774315
Title: Molecular Endotypes of Chronic Idiopathic Urticaria
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-0850
Record Dates: First submitted 2021-02-16; First posted 2021-03-01 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Chronic Urticaria, Idiopathic
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Omalizumab (Experimental)
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — omalizumab 300mg SQ every 4 weeks as part of standard of care

SUMMARY:
This study plans to learn more about why some people with Chronic Idiopathic Urticaria (CIU) respond to treatment with omalizumab (Xolair). It will test people before they receive treatment with omalizumab as part of standard of care, to see if there are differences in their blood and skin that can predict who responds to treatment.

ELIGIBILITY:
Inclusion Criteria:

* CIU as defined as frequent urticarial lesions for ≥ 6 weeks
* Symptoms not controlled with standard dose antihistamines (loratadine 10mg daily, desloratadine 5mg daily, fexofenadine 180mg daily, cetirizine 10mg daily, or levocetirizine 5mg daily)
* Planned initiation of treatment with omalizumab (Xolair) as part of standard of care for antihistamine-refractory urticaria

Exclusion Criteria:

* Use of immunomodulatory drugs in the past 1 month prior to beginning the study
* Use of systemic steroids in the past 1 month prior to beginning the study
* Use of omalizumab in the past 3 months prior to beginning the study
* Use of any investigational agent in the past 30 days
* Untreated intercurrent illness
* Severe Asthma
* Primary diagnosis of flushing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Responders | Week 16
  The number of participants who meet the definition of "Responder" to omalizumab. "Responders" are defined as having a UAS7 of 6 or less after 16 weeks of treatment.

SECONDARY OUTCOMES:
Baseline expression of innate immune markers | Baseline
  Baseline expression of innate immune markers in peripheral blood between eventual responders and nonresponders to omalizumab. 5 significant markers will be reported. Results will be stratified between groups determined by the pre-specified arms and by the classification of participants as responders versus non-responders to omalizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Stitt, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No